CLINICAL TRIAL: NCT02767375
Title: Hepatic Arterial Infusion Chemotherapy as Adjuvant Treatment in the Prevention of Recurrence of Hepatocellular Carcinoma(HCC): A Prospective Randomized Controlled Clinical Trial
Brief Title: Hepatic Arterial Infusion Chemotherapy(HAIC) for Hepatoma After Resection
Acronym: HAICAT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Baocai Xing, The chief of Department of Hepatobiliary Pancreatic Surgery Ward, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BeijingCancerH
Record Dates: First submitted 2016-04-03; First posted 2016-05-10 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Hepatic arterial infusion chemotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HAIC treatment group (Active Comparator): HAIC treatment after resection Intervention: Drug: Oxaliplatin, 5-fluorouracil (5-FU) Procedure/Surgery: Hepatic arterial catheter implantation
  Interventions: Drug: Oxaliplatin(OXA), 5-fluorouracil (5-FU); Procedure: Hepatic arterial catheter implantation
- No HAIC treatment group (No Intervention): Best support care and follow up

INTERVENTIONS:
Drug: Oxaliplatin(OXA), 5-fluorouracil (5-FU) — for the HAIC treatment group OXA 85mg/m2, d1，0-4h 5-FU 1500mg/m2 d1, 4-24h 24 hours in d1 & 2 , IA，q4-6 Weeks
  Other Names: OXA,5-FU
  Arms: HAIC treatment group
Procedure: Hepatic arterial catheter implantation — for the the HAIC treatment group: Hepatic arterial catheter implantation for HAIC
  Other Names: HAIC
  Arms: HAIC treatment group

SUMMARY:
To study if the addition of HAIC following complete removal of early stage liver cancer of HCC will prevent or delay the recurrence of the disease. Half of the participant will receive two cycles of the HAIC after the hepatectomy, while the other half will return to the baseline surveillance schedule.

DETAILED DESCRIPTION:
The high incidence of HCC recurrence following liver resection is a serious issue. The recurrent rate is as high as 50-60% at 3 years and 70-100% at 5 years.

So to reduce the recurrence rate of HCC, some interventions had been tried in clinic, including transarterial chemoembolization (TACE), immunotherapy, and interferon treatment etc. But few of these adjuvant therapies had been proved effective and the long term efficacy and clinical application remained further explored.

HAIC had been prove to be effective adjuvant treatment in patients with liver metastasis of colorectal cancers in randomized controlled trials and meta-analysis, but the role of adjuvant HAIC after liver resection is controversial. The results getting from different randomized control trials varied significantly because of the bias of patient selection, different study design，the small size of sample, different drug used in chemotherapy and lack of proper stratification,so a big sample size, well patients selected and well designed randomized controlled trial is needed to further confirm the role of the postoperative HAIC.

Patients with HCC who received curative liver resection (R0) were randomly assigned 1:1 by the doctors to receive no adjuvant HAIC(control group) or HAIC (treatment group). All patients in the treatment group will receive 2 cycles of adjuvant HAIC within 3 months after liver resection. The outcomes of patients were evaluated during the 5-years follow up.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Informed consent Confirmation of diagnosis of HCC: For subjects undergoing surgical resection histological confirmation is mandatory (a post surgery pathology report is required for both histological confirmation and risk stratification).
* After qualifying at the time of scanning, by independent radiology review diagnosed CR (no residual tumor deposit radical therapy Assess their level of risk of disease recurrence by tumor characteristics as moderate or high risk
* Subjects who have undergone surgical resection for treatment of HCC with curative intent within 4 months from staging to potentially curative treatment.
* At least 3 weeks (21 days) but not more than 7 weeks (49 days), from resection course, to CT/MRI scan date. A timeframe of 4 weeks after surgical resection is recommended.
* Male or female subjects ≥ 18 years of age Confirmation of complete response(CR)- (absence of residual tumor after curative treatment), on the eligibility scan by independent radiological review.
* For subjects undergoing surgical resection pathology proven complete removal of tumor. Intermediate or High Risk of recurrence as assessed by tumor characteristics.
* Child-Pugh score 5 -7 points. A Child-Pugh score of 7 points is allowed only in the absence of ascites.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0.
* Adequate bone marrow, liver and renal function as assessed by central lab by means of the following laboratory requirements from samples within 14 days prior to randomization: Alpha fetoprotein ≤ 400 ng/mL
* Women of childbearing potential must have a negative serum pregnancy test performed within 14 days prior to the start of treatment (assessed centrally).

Exclusion Criteria:

* Recurrent HCC Child-Pugh score 7 points with presence of ascites.
* The following tumor characteristics: Low risk of recurrence after curative treatment defined as any of the following: for local ablation patients: single lesions ≤ 2 cm for surgical resection patients: single lesions ≤ 2 cm without microscopic vascular invasion, without tumor satellites and histologically well differentiated. ≥ 3 lesions or 2-3 lesions of which any are ≥ 3 cm in size (largest diameter, unidimensional measurement) prior curative treatment (surgical resection or local ablation) single lesion ≥ 5 cm (largest diameter, unidimensional measurement) in size prior local ablation.
* Macrovascular invasion Extrahepatic spread (including regional lymph nodes and invasion into adjacent structures)
* History of cardiovascular disease:
* History of HIV infection Active clinically serious infections (≥ grade 2 NCI-CTCAE version 3.0)
* Subjects with seizure disorder requiring medication (such as steroids or anti-epileptics)
* History of organ allograft Subjects with evidence or history of bleeding diathesis
* Subjects undergoing renal dialysis
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated ≥ 3 years prior to study entry as defined by the signing of informed consent.
* Uncontrolled ascites (defined as not easily controlled with diuretic treatment)
* Encephalopathy History of GI bleeding within 30 days of randomization.
* Subjects with a history of esophageal varices bleeding which has not been followed by effective therapy and/or treatment to prevent bleeding recurrence.
* Prior anti cancer therapy for treatment of HCC (including sorafenib or any other molecular therapy) is excluded.
* Major surgery within 4 weeks of start of study as defined by the signing of informed consent, except for surgical resection or local ablation of HCC.
* Autologous bone marrow transplant or stem cell rescue within 4 months of study entry as defined by the signing of informed consent.
* Use of biologic response modifiers, such as colony stimulating factor(G-CSF), within 3 week of study entry, as defined by the signing of informed consent.
* Investigational drug therapy outside of this trial during or within 4 weeks of study entry, as defined by the signing of informed consent.
* Pregnant or breast-feeding subjects.
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results
* Known or suspected allergy to contrast media for angiography.
* Any condition that is unstable or could jeopardize the safety of the subject and their compliance in the study
* This applies to subjects with severe obstruction of the upper GI tract that require gavage.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free Survival | approximately 70 months from first patient first visit

SECONDARY OUTCOMES:
Time to recurrence | approximately 60 months from first patient first visit
Overall survival | approximately 60 months from first patient first visit
Visual Analog Score for pain | approximately 60 months from first patient first visit
Physicians Global Assessment to measure quality of life | approximately 60 months from first patient first visit
Number of Participants With Abnormal Laboratory Values | approximately 60 months from first patient first visit
Adverse Events That Are Related to Treatment | approximately 60 months from first patient first visit

CONTACTS AND LOCATIONS:
Overall Officials: Baocai Xing, Doctor, Study Director — 1st Department of HBP Surgery.Beijing Cancer Hospital; Xu Zhu, Doctor, Study Director — Interventional therapy department of Beijing Cancer Hospital
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clinical Practice Guidelines for Hepatocellular Carcinoma Differ between Japan, United States, and Europe. Liver Cancer. 2015 Mar;4(2):85-95. doi: 10.1159/000367730. No abstract available. PMID 26020031
- [Background] Qi X, Liu L, Wang D, Li H, Su C, Guo X. Hepatic resection alone versus in combination with pre- and post-operative transarterial chemoembolization for the treatment of hepatocellular carcinoma: A systematic review and meta-analysis. Oncotarget. 2015 Nov 3;6(34):36838-59. doi: 10.18632/oncotarget.5426. PMID 26451613
- [Background] Lee JH, Lee Y, Lee M, Heo MK, Song JS, Kim KH, Lee H, Yi NJ, Lee KW, Suh KS, Bae YS, Kim YJ. A phase I/IIa study of adjuvant immunotherapy with tumour antigen-pulsed dendritic cells in patients with hepatocellular carcinoma. Br J Cancer. 2015 Dec 22;113(12):1666-76. doi: 10.1038/bjc.2015.430. Epub 2015 Dec 10. PMID 26657650
- [Background] Zhong JH, Li H, Li LQ, You XM, Zhang Y, Zhao YN, Liu JY, Xiang BD, Wu GB. Adjuvant therapy options following curative treatment of hepatocellular carcinoma: a systematic review of randomized trials. Eur J Surg Oncol. 2012 Apr;38(4):286-95. doi: 10.1016/j.ejso.2012.01.006. Epub 2012 Jan 24. PMID 22281155
- [Background] Kumamoto T, Tanaka K, Matsuo K, Takeda K, Nojiri K, Mori R, Taniguchi K, Matsuyama R, Ueda M, Akiyama H, Ichikawa Y, Ota M, Endo I. Adjuvant hepatic arterial infusion chemotherapy with 5-Fluorouracil and interferon after curative resection of hepatocellular carcinoma: a preliminary report. Anticancer Res. 2013 Dec;33(12):5585-90. PMID 24324102
- [Background] Tung-Ping Poon R, Fan ST, Wong J. Risk factors, prevention, and management of postoperative recurrence after resection of hepatocellular carcinoma. Ann Surg. 2000 Jul;232(1):10-24. doi: 10.1097/00000658-200007000-00003. PMID 10862190
- [Background] Nitta H, Beppu T, Imai K, Hayashi H, Chikamoto A, Baba H. Adjuvant hepatic arterial infusion chemotherapy after hepatic resection of hepatocellular carcinoma with macroscopic vascular invasion. World J Surg. 2013 May;37(5):1034-42. doi: 10.1007/s00268-013-1957-1. PMID 23435678
- [Background] Nagano H. Treatment of advanced hepatocellular carcinoma: intraarterial infusion chemotherapy combined with interferon. Oncology. 2010 Jul;78 Suppl 1:142-7. doi: 10.1159/000315243. Epub 2010 Jul 8. PMID 20616597
- [Background] Song MJ. Hepatic artery infusion chemotherapy for advanced hepatocellular carcinoma. World J Gastroenterol. 2015 Apr 7;21(13):3843-9. doi: 10.3748/wjg.v21.i13.3843. PMID 25852268
- [Background] Shiozawa K, Watanabe M, Ikehara T, Kogame M, Matsui T, Okano N, Kikuchi Y, Nagai H, Ishii K, Makino H, Igarashi Y, Sumino Y. Comparison of Sorafenib and Hepatic Arterial Infusion Chemotherapy for Advanced Hepatocellular Carcinoma: A Propensity Score Matching Study. Hepatogastroenterology. 2014 Jun;61(132):885-91. PMID 26158136
- [Background] Bruix J, Takayama T, Mazzaferro V, Chau GY, Yang J, Kudo M, Cai J, Poon RT, Han KH, Tak WY, Lee HC, Song T, Roayaie S, Bolondi L, Lee KS, Makuuchi M, Souza F, Berre MA, Meinhardt G, Llovet JM; STORM investigators. Adjuvant sorafenib for hepatocellular carcinoma after resection or ablation (STORM): a phase 3, randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2015 Oct;16(13):1344-54. doi: 10.1016/S1470-2045(15)00198-9. Epub 2015 Sep 8. PMID 26361969
- [Result] Korean Liver Cancer Study Group (KLCSG); National Cancer Center, Korea (NCC). 2014 Korean Liver Cancer Study Group-National Cancer Center Korea practice guideline for the management of hepatocellular carcinoma. Korean J Radiol. 2015 May-Jun;16(3):465-522. doi: 10.3348/kjr.2015.16.3.465. Epub 2015 May 13. PMID 25995680